CLINICAL TRIAL: NCT02265003
Title: Red Blood Cells as a Reflection of Endothelial Function in Old Age
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator Prof. Dr. Malte Kelm, Heinrich-Heine University, Duesseldorf
Other Study IDs: Anaemie; 14-016 (Other: CTSU)
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Red Blood Cells; Endothelial Function; Nitric Oxide Pool in Red Blood Cells and Blood Plasma
Keywords: red blood cells; endothelial function; nitric oxide pool in red blood cells; nitric oxide poll in blood plasma; nitric oxide synthase III - expression; oxidative status; nitric oxide signalling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy young age: Healthy subjects in age of 18-35 years, without cardiac dysrhythmia, hypertension, diabetes mellitus, acute inflammations and terminal kidney disease
- Healthy middle age: Healthy subjects in age of 35-45 years, without cardiac dysrhythmia, hypertension, diabetes mellitus, acute inflammations and terminal kidney disease
- Healthy old: Healthy subjects in age of >70 years, without cardiac dysrhythmia, hypertension, diabetes mellitus, acute inflammations and terminal kidney disease
- Patients: Patients with atherosclerosis

SUMMARY:
The aim of this study is to find out, how far red blood cells reflect age-depended changes in endothelial function.

DETAILED DESCRIPTION:
It will be investigated with determination of endothelial function (measured as flow-mediated vasodilation) and of circulated nitric oxid-pool in red blood cells and in blood plasma, how far red blood cells reflect age-depended changes in endothelial function.

ELIGIBILITY:
Groups 1-3:

Inclusion Criteria:

* healthy subjects
* informed consent

Exclusion Criteria:

* hypertension (blood pressure ≥140/90 mmHg),
* hypercholesterolemia (LDL ≥250 mg/dl, HDL ≤45 mg/dl),
* diabetes mellitus (fasting plasma glucose ≥128 mg/dl)
* acute inflammation (CRP >0.5 mg/dl)
* malignant diseases
* heart failure (NYHA III-IV)
* arrhythmia of high degree
* acute or terminated kidney disease
* cardiovascular diseases ( cardiac artery disease, peripheral vascular disease and cerebrovascular diseases)
* anemia
* pregnancy

Group 4 :

Inclusion Criteria:

* angiographical signs of apparent atherosclerosis (cardiac artery disease or peripheral vascular disease or degenerative valvular heart disease)
* informed consent

Exclusion Criteria:

* Hypertension (blood pressure ≥140/90 mmHg),
* Hypercholesterolemia (LDL ≥250 mg/dl, HDL ≤45 mg/dl),
* Diabetes mellitus (fasting plasma glucose ≥128 mg/dl)
* acute inflammation (CRP >0.5 mg/dl)
* malignant diseases
* heart failure (NYHA III-IV)
* arrhythmia of high degree
* acute or terminated kidney disease
* cardiovascular diseases ( cardiac artery disease, peripheral vascular disease and cerebrovascular diseases)
* anemia
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 4 groups:
  * healthy young aged 18-35 years (30 subjects)
  * healthy middel aged 35-45 years (30 subjects)
  * healthy old aged > 70 years (30 subjects)
  * patients (50 subjects)
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2012-07; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Determination of endothelial function | baseline
  measured as flow-mediated vasodilation

SECONDARY OUTCOMES:
Determination of nitric oxide(NO)-pool in red blood cells and blood plasma | baseline
Determination of erythrocytes parameter | baseline
  It will be determinated: oxidative status, signalling of nitric oxide, function, creation, amount and aging of red blood cells, cell-to-cell-interaction, microRNA and inflammation
Cardiovascular Parameter | baseline
  It will be determinated: hemodynamic, microcirculation and physicomechanic

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof. MD, Principal Investigator — Department of Cardiology, Pneumology and Angiology, University Hospital Duesseldorf
Locations (1):
- University Hospital Duesseldorf, Düsseldorf, Germany